CLINICAL TRIAL: NCT06233435
Title: Comparison of Modified Post-Anesthetic Discharge Scoring System (PADSS) Between 6 and 24 Hours in Patients Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Niruji Saengsomsuan, Anesthesiology, Thammasat University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-AN-2-179/66
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-05

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PADSS at 6 hours (Other)
  Interventions: Behavioral: PADSS
- PADSS at 24 hours (Other)
  Interventions: Behavioral: PADSS

INTERVENTIONS:
Behavioral: PADSS — Observe PADSS after total knee arthroplasty at 6 and 24 hours

SUMMARY:
This study is a prospective study which compares of Modified Post-Anesthetic Discharge Scoring System (PADSS) between 6 and 24 hours in patients undergoing total knee arthroplasty in Thammasat University hospital, Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing total knee arthroplasty (one side) under spinal block with adductor canal block
* 18-85 years old
* American Society of Anesthesiologist physical status classification I-III

Exclusion Criteria:

* Allergy to local anesthetic drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Comparison of Modified Post-Anesthetic Discharge Scoring System (PADSS) Between 6 and 24 Hours in Patients Undergoing Total Knee Arthroplasty | at 6 and 24 hours after total knee arthroplasty

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University hospital, Pathum Thani, Klong Luang, Thailand

IPD SHARING:
Plan to Share IPD: No